CLINICAL TRIAL: NCT04879641
Title: Optimizing Cognitive-behavioral Therapy for Social Anxiety Disorder Using the Factorial Design: What Works Best and How Does it Work (OPTIMIZE)
Brief Title: Optimizing Cognitive-behavioral Therapy for Social Anxiety Disorder Using the Factorial Design
Acronym: OPTIMIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: OPTIMIZE_TRIAL
Record Dates: First submitted 2021-04-09; First posted 2021-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Social Anxiety Disorder (Social Phobia)
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: The study is a single-center, factorial trial with four experimental factors (treatment components, i.e., psychoeducation, cognitive restructuring, attention training, and exposure) each evaluated at two levels (presence vs. absence) resulting in 16 treatment conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- 1_Waiting List control (No Intervention): Randomized participants will only get the full intervention after study completion period (6 months since the randomization)
- 2_Exposure only (Experimental): Randomized participants will only get the Exposure component
  Interventions: Behavioral: Exposure
- 3_Attention Training only (Experimental): Randomized participants will only get the Attention Training component
  Interventions: Behavioral: Attention Training
- 4_Exposure + Attention Training (Experimental): Randomized participants will get Exposure + Attention Training components
  Interventions: Behavioral: Exposure; Behavioral: Attention Training
- 5_Cognitive Restructuring only (Experimental): Randomized participants will only get the Cognitive Restructuring component
  Interventions: Behavioral: Cognitive Restructuring
- 6_Cognitive Restructuring + Exposure (Experimental): Randomized participants will get Cognitive Restructuring + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Cognitive Restructuring
- 7_Cognitive Restructuring + Attention Training (Experimental): Randomized participants will get Cognitive Restructuring + Attention Training components
  Interventions: Behavioral: Attention Training; Behavioral: Cognitive Restructuring
- 8_Cognitive Restructuring + Attention Training + Exposure (Experimental): Randomized participants will get Cognitive Restructuring + Attention Training + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Attention Training; Behavioral: Cognitive Restructuring
- 9_Psychoeducation only (Experimental): Randomized participants will only get the Psychoeducation component
  Interventions: Behavioral: Psychoeducation
- 10_Psychoeducation + Exposure (Experimental): Randomized participants will get the Psychoeducation + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Psychoeducation
- 11_Psychoeducation + Attention Training (Experimental): Randomized participants will get the Psychoeducation + Attention Training components
  Interventions: Behavioral: Attention Training; Behavioral: Psychoeducation
- 12_Psychoeducation + Attention Training + Exposure (Experimental): Randomized participants will get the Psychoeducation + Attention Training + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Attention Training; Behavioral: Psychoeducation
- 13_Psychoeducation + Cognitive Restructuring (Experimental): Randomized participants will get the Psychoeducation + Cognitive Restructuring components
  Interventions: Behavioral: Cognitive Restructuring; Behavioral: Psychoeducation
- 14_Psychoeducation + Cognitive Restructuring + Exposure (Experimental): Randomized participants will get the Psychoeducation + Cognitive Restructuring + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Cognitive Restructuring; Behavioral: Psychoeducation
- 15_Psychoeducation + Cognitive Restructuring + Attention Training (Experimental): Randomized participants will get the Psychoeducation + Cognitive Restructuring + Attention Training components
  Interventions: Behavioral: Attention Training; Behavioral: Cognitive Restructuring; Behavioral: Psychoeducation
- 16_full version (Psychoeducation + Cognitive Restructuring + Attention Training + Exposure) (Experimental): Randomized participants will get the Psychoeducation + Cognitive Restructuring + Attention Training + Exposure components
  Interventions: Behavioral: Exposure; Behavioral: Attention Training; Behavioral: Cognitive Restructuring; Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Exposure — Participants are instructed to plan and track in vivo exposures using an exposure diary. Participants are also instructed to reduce safety behaviors, which are overt or covert acts such as avoiding eye contact or rehearsing sentences to prevent a feared outcome.
  Arms: 10_Psychoeducation + Exposure; 12_Psychoeducation + Attention Training + Exposure; 14_Psychoeducation + Cognitive Restructuring + Exposure; 16_full version (Psychoeducation + Cognitive Restructuring + Attention Training + Exposure); 2_Exposure only; 4_Exposure + Attention Training; 6_Cognitive Restructuring + Exposure; 8_Cognitive Restructuring + Attention Training + Exposure
Behavioral: Attention Training — Participants are trained to reduce self-focused and biased attention. Various audio exercises are introduced in which participants learn to intentionally direct the attention away from themselves (i.e., less private self-consciousness), and to be less alert to potentially dangerous external social stimuli (i.e., less public self-consciousness).
  Arms: 11_Psychoeducation + Attention Training; 12_Psychoeducation + Attention Training + Exposure; 15_Psychoeducation + Cognitive Restructuring + Attention Training; 16_full version (Psychoeducation + Cognitive Restructuring + Attention Training + Exposure); 3_Attention Training only; 4_Exposure + Attention Training; 7_Cognitive Restructuring + Attention Training; 8_Cognitive Restructuring + Attention Training + Exposure
Behavioral: Cognitive Restructuring — Participants are instructed to identify and modify dysfunctional and negatively biased assumptions. It includes a thought diary to track negative beliefs in daily routine, alongside with exercises to formulate helpful and adaptive thoughts.
  Arms: 13_Psychoeducation + Cognitive Restructuring; 14_Psychoeducation + Cognitive Restructuring + Exposure; 15_Psychoeducation + Cognitive Restructuring + Attention Training; 16_full version (Psychoeducation + Cognitive Restructuring + Attention Training + Exposure); 5_Cognitive Restructuring only; 6_Cognitive Restructuring + Exposure; 7_Cognitive Restructuring + Attention Training; 8_Cognitive Restructuring + Attention Training + Exposure
Behavioral: Psychoeducation — Participants are delivered detailed evidence-based information on SAD with a focus on maintaining processes (e.g., the vicious circle of negative thoughts and emotions, cognitions, and behaviors associated with the maintenance of SAD). Based on the information provided, participants are encouraged to develop an individual model of their social anxiety symptoms.
  Arms: 10_Psychoeducation + Exposure; 11_Psychoeducation + Attention Training; 12_Psychoeducation + Attention Training + Exposure; 13_Psychoeducation + Cognitive Restructuring; 14_Psychoeducation + Cognitive Restructuring + Exposure; 15_Psychoeducation + Cognitive Restructuring + Attention Training; 16_full version (Psychoeducation + Cognitive Restructuring + Attention Training + Exposure); 9_Psychoeducation only

SUMMARY:
Social Anxiety Disorder (SAD) is characterized by a marked fear of negative evaluation in social situations. It is the third most common psychiatric disorder and highly disabling (American Psychiatric Association, 2000). Although effective treatments such as cognitive-behavioral therapy (CBT) are available, most individuals suffering from SAD do not seek and eventually find help, and even in the best available treatments, remission rates are below 50%. The overall aim of the project is to better understand and improve the efficacy of Internet-based CBT (ICBT) that has shown to be efficacious in many trials and that provide broad and low-threshold access to empirically supported treatments. Specifically the objectives of the study are:

1. to investigate the active ingredients of ICBT for SAD by testing the main effects and interactions for the four main treatment components (i.e., psychoeducation, cognitive restructuring, attention training, and exposure);
2. to investigate the effects of each treatment component on hypothesized change mechanisms, and to explore whether and which change mechanisms mediate the effect of the treatment components on symptom reduction.
3. to investigate whether the specific mechanisms mediate the effect of the treatment components on primary and secondary outcomes.

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is characterized by a marked fear of negative evaluation in social situations. It is the third most common psychiatric disorder and highly disabling. Although effective treatments such as cognitive-behavioral therapy (CBT) are available, most individuals suffering from SAD do not seek and eventually find help, and even in the best available treatments, remission rates are below 50%. The overall aim of the project is to improve the efficacy of Internet-based CBT (ICBT) that has shown to be efficacious in many trials and that provide broad and low-threshold access to empirically supported treatments. Specifically, the objectives of the study are:

1. to investigate the active ingredients of ICBT for SAD by testing the main effects and interactions for the four main treatment components (i.e., psychoeducation, cognitive restructuring, attention training, and exposure);
2. to investigate the effects of each treatment component on hypothesized change mechanisms (change of the knowledge of SAD, change on negative social cognitions, changes on self-focused attention, changes on social avoidance and use of safety behaviors), and to explore whether and which change mechanisms mediate the effect of the treatment components on symptom reduction.
3. to investigate whether the specific mechanisms mediate the effect of the treatment components on primary and secondary outcomes.

The study is a single-center, factorial trial with four experimental factors (treatment components, i.e., psychoeducation, cognitive restructuring, attention training, and exposure) each evaluated at two levels (presence vs. absence) resulting in 16 conditions.

Recruitment: Participants will be recruited using reports in newspapers, through internet forums, social media (e.g., Facebook), and via our website (https://www.online-therapy.ch/) in German-speaking countries.

Sampling: After checking the inclusion criteria, participants will be randomized with equal probability to one of the 16 conditions. The random allocation will be unknown to the investigators. In order to keep the sample sizes of the 16 conditions similar, the allocation list will be made using randomly permuted blocks. A total of 464 participants with a Diagnostic and Statistical Manual of Mental Disorders diagnosis of SAD will be included, with 29 patients being assigned to each of the 16 conditions.

Assessment procedures: The primary outcome measure is change in symptoms of SAD at post-treatment, i.e., after 8 weeks. Secondary outcomes include sustaining change at follow up (6 months after baseline), changes in depressive symptoms, changes in general anxiety symptoms, changes in quality of life, adherence to treatment, treatment satisfaction, negative effects and changes of diagnosis of SAD. Furthermore, the hypothesized change mechanisms (change of the knowledge of SAD, change on negative social cognitions, changes in self-focused attention, changes in social avoidance and use of safety behaviors) will be assessed. Self-report measures are taken at pre-treatment (baseline), after 4 weeks (mid-treatment), after 8 weeks (post-treatment), and at 6 months after randomization (follow-up). Besides the self-report measures, a diagnostic interview will be conducted by phone at pre-treatment, eight weeks (posttreatment), and six months (follow-up). The structured M.I.N.I. Interview will be used. The interviews will be administered by advanced Master students in clinical psychology and psychotherapy supervised by the study team. Interrater reliability will be assessed on a subset of the cases.

Treatment: The internet-based self-help program ("Shyne", https://selfhelp1.psy.unibe.ch/shyne/) is based on the well-established cognitive-behavioral treatment of social anxiety by Clark and Wells and has been proven efficacious in previous studies. Shyne is accessed through a secure website, with each participant having a password-protected account. It consists of the following four treatment components: (1) psychoeducation (knowledge about SAD and its treatment); (2) cognitive restructuring (challenging dysfunctional social cognitions); (3) attention training (decrease of self-focused attention); and (4) exposure (decrease of avoidance of feared situations and safety behaviors). These treatment components will be offered in 16 different combinations.

Data analysis: Primary analyses will be conducted on the Intention-To-Treat (ITT) sample (i.e., all randomized participants). The analyses are carried out on the basis of the intention-to-treat (ITT) approach using linear mixed models. In addition, but only secondary, completers analysis will be carried out. In order to test for main and interaction effects of treatment components on outcomes and change mechanisms across the time points of assessment, linear mixed models Analysis of Variance (ANOVA) or latent growth curve modelling will be used. Main effects and interactions will be based on aggregates across experimental conditions. Sensitivity analyses will explore the impact of the imputation of missing values. For binary outcome data (i.e., SAD diagnosis), a logistic regression model will be used. Furthermore, mediation analyses will be used to determine whether the hypothesized change mechanisms mediate the effect of the treatment components on primary and secondary outcomes. The mediation will be tested using an approach that allows multiple mediators in one model. In addition, potential moderation of the treatment components by various measured variables such as comorbid disorder, medication, the severity of SAD, age and sex will be investigated. Reporting will follow CONSORT E-Health standards.

ELIGIBILITY:
Inclusion Criteria:

* 1. read the study information and sign informed consent;
* 2. are 18 years or older;
* 3. have access to the Internet, to a smartphone, PC or tablet;
* 4. have sufficient knowledge of German;
* 5. exceed predefined cut-off scores on one of the social anxiety measures (22 points on the Social Phobia Scale or 33 points on the Social Interaction Anxiety Scale; SPS & SIAS);
* 6. fulfil the diagnostic criteria of SAD according to the diagnostic telephone interview (the presence of other disorders does not result in exclusion if SAD is the primary diagnosis)
* 7. in the case of taking psychiatric medication, the treatment is stabilized (over one month)

Exclusion Criteria:

* 1. they score 2 or higher on the suicide item of the PHQ-9 (Spitzer, 1999) or with active suicidal plans in the diagnostic telephone interview.
* 2. they have other comorbid psychiatric conditions that might be the main focus of clinical attention (e.g., psychotic symptoms, bipolar disorder, or other severe disorder)
* 3. they undergo another psychological treatment at the beginning of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change on social anxiety symptoms at post-treatment | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline)
  Composite endpoint. Social anxiety symptoms are measured as the combined score of the Social Phobia Scale and the Social Interaction Anxiety Scale (SPS & SIAS; Mattick & Clarke, 1998). These instruments are complementary and used as one single measurement. They assess the fear of being judged by others during daily activities (SPS) and more general fears in social interaction (SIAS). The combined scale consists of 40 items and scores range from 0 (no social anxiety symptoms) to 160 (severe social anxiety symptoms).

SECONDARY OUTCOMES:
Change on social anxiety symptoms at follow-up | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Social anxiety symptoms are measured as the combined score of the Social Phobia Scale and the Social Interaction Anxiety Scale (SPS & SIAS; Mattick & Clarke, 1998). These instruments are complementary and used as one measurement. They assess the fear of being judged by others during daily activities (SPS) and more general fears in social interaction (SIAS). The combined scale consists of 40 items and scores range from 0 (no social anxiety symptoms) to 160 (severe social anxiety symptoms).
Change on the severity of depressive symptoms | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Depressive symptoms will be measured by the Patient Health Questionnaire (PHQ-9; Spitzer et al., 1999). Scores range from 0 (no depressive symptoms) to 27 (severe depressive symptoms).
Change on the severity of general anxiety symptoms | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Severity of anxiety symptoms will be measured by the Generalized Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006). Scores range from 0 (no general anxiety symptoms) to 21 (severe general anxiety symptoms)
Change on quality of life | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Quality of life will be measured by the Short-Form Health Survey-12 (SF-12; Ware et al., 1996). Scores range from 12 (high quality of life) to 53 (poor quality of life).
Level of satisfaction with the treatment | Post-treatment (8 weeks after baseline)
  Treatment satisfaction will be measured by the Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982), adapted to internet-based interventions. Scores range from 0 (not satisfied at all) to 24 (extremely satisfied).
Negative effects of the treatment | Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Adverse effects on social, intrapersonal or work-related situations and whether they are attributed to the intervention will be measured on the 15 items Negative Effects of the Treatment scale (INEP; Ladwig et al., 2014). The scores range from - 39 (worse) to +18 (best), in which negative values indicate negative effects of the intervention
Change on the diagnosis of social anxiety disorder | Baseline, Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Diagnosis of social anxiety disorder will be assessed with M.I.N.I International Neuropsychiatric Interview for DSM-IV 6.0.0 (M.I.N.I; Sheehan et al., 1998). Possible diagnoses are absence or presence of SAD, current or past, generalized or specific, primary diagnosis (yes or no)

OTHER OUTCOMES:
Change on the knowledge of social anxiety disorder | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Basic knowledge around the condition of SAD and its treatment will be assessed with the Knowledge of SAD test (KSAD; Andersson, et al., 2012). The scores range from 0 to 33, the higher the score, more knowledge about SAD
Change on negative social cognitions | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Typical negative social cognitions of socially anxious individuals will be assessed with the Social Cognitions Questionnaire (SCQ; Wells et al., 1993). Scores range from 22 to 110, and higher scores mean more negative social cognitions
Change on self-focused attention (or self-consciousness) | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Self-focused attention (or self-consciousness) in two dimensions (private self-consciousness and public self-consciousness) will be assessed with the Self-Consciousness Scale (SCS; Fenigstein et al., 1975). Scores range from 27 to 135. Higher scores means more self-focused attention.
Change on social avoidance and intensity of distress facing social situations | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  Social avoidance and the intensity of fear/anxiety facing social situations will be assessed with the Liebowitz Social Anxiety Scale, self-report (LSAS-SR; Baker et al., 2002). Scores range from 0 to 144. Higher scores mean more avoidance of and fear in social situations
Change on the use of safety behaviors in social situations | Baseline, Mid-treatment (4 weeks after baseline), Post-treatment (8 weeks after baseline), Follow-up (6 months after baseline)
  The use of safety behaviors in social situations will be assessed with the Social Behaviors Questionnaire (SBQ; Clark et al., 1995). Scores range from 0 to 81. Higher scores mean more use of safety behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Thomas T Berger, Prof., Principal Investigator — University Bern, Clinical Psychology and Psychotherapy Department
Locations (1):
- Clinical Psychology and Psychotherapy Department, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Berger T, Hohl E, Caspar F. Internet-based treatment for social phobia: a randomized controlled trial. J Clin Psychol. 2009 Oct;65(10):1021-35. doi: 10.1002/jclp.20603. PMID 19437505
- [Background] Schulz A, Stolz T, Vincent A, Krieger T, Andersson G, Berger T. A sorrow shared is a sorrow halved? A three-arm randomized controlled trial comparing internet-based clinician-guided individual versus group treatment for social anxiety disorder. Behav Res Ther. 2016 Sep;84:14-26. doi: 10.1016/j.brat.2016.07.001. Epub 2016 Jul 7. PMID 27423374
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Andersson G, Carlbring P, Furmark T; S. O. F. I. E. Research Group. Therapist experience and knowledge acquisition in internet-delivered CBT for social anxiety disorder: a randomized controlled trial. PLoS One. 2012;7(5):e37411. doi: 10.1371/journal.pone.0037411. Epub 2012 May 23. PMID 22649526
- [Background] Watson D, Friend R. Measurement of social-evaluative anxiety. J Consult Clin Psychol. 1969 Aug;33(4):448-57. doi: 10.1037/h0027806. No abstract available. PMID 5810590
- [Background] American Psychiatric Association. (2000). DSM-IV: Diagnostic and Statistical Manual of Mental Disorders (4th). Author.
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. In R. G. Heimberg, M. R. Liebowitz, D. Hope, & F. Schneider (Eds.), Social Phobia: Diagnosis, Assessment, and Treatment (pp. 69-93). Guilford Press.
- [Background] Ladwig, I., Rief, W., & Nestoriuc, Y. (2014). What Are the Risks and Side Effects of Psychotherapy? - Development of an Inventory for the Assessment of Negative Effects of Psychotherapy (INEP). Verhaltenstherapie, 24(4), 252-263. https://doi.org/0.1159/000367928
- [Background] Wells, A., Stopa, L., & Clark, D. M. (1993). The social cognitions questionnaire. Unpublished, Department of Psychiatry, University of Oxford, Warnerford Hospital, Oxford, UK.
- [Background] Fenigstein, A., Scheier, M. F., & Buss, A. H. (1975). Public and private self-consciousness: Assessment and theory. Journal of Consulting and Clinical Psychology, 43(4), 522-527. https://doi.org/10.1037/h0076760
- [Background] Clark, D. M., Wells, A., Salkoviskis, P., & Hackmann, A. (1995). Social behaviour questionnaire [Unpublished Manuscript].
- [Derived] Sipka D, Lopes R, Krieger T, Klein JP, Berger T. Active Components in Internet-Based Cognitive-Behavioral Therapy for Social Anxiety Disorder: A Randomized Full Factorial Trial. Psychother Psychosom. 2025;94(1):40-59. doi: 10.1159/000542425. Epub 2025 Jan 10. PMID 39799943
- [Derived] Lopes RCT, Sipka D, Krieger T, Klein JP, Berger T. Optimizing cognitive-behavioral therapy for social anxiety disorder and understanding the mechanisms of change: Study protocol for a randomized factorial trial. Internet Interv. 2021 Nov 10;26:100480. doi: 10.1016/j.invent.2021.100480. eCollection 2021 Dec. PMID 34824982
- See also: The guided internet-based program Shyne, which will be the studied treatment (requires password) — https://selfhelp1.psy.unibe.ch/shyne/